CLINICAL TRIAL: NCT04312711
Title: To Assess the Value of 3D Time-of-Flight Magnetic Resonance Angiography in Hemodialysis Patients With Occlusive Disease in Arteriovenous Fistula
Brief Title: 3D Time-of-Flight Magnetic Resonance Angiography in Hemodialysis Patients With Arteriovenous Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Shanghai 6th People's Hospital
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Magnetic Resonance Angiography; Hemodialysis; Arteriovenous Fistula Stenosis
MeSH Terms: interventions — Ultrasonography; Angiography, Digital Subtraction

STUDY DESIGN:
Intervention Model Description: All participants will receive three-dimensional time-of-flight magnetic resonance angiography (3D-TOF-MRA) and ultrasound to detect the stenosis degree of AVF.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): All participants received 3D-TOF-MRA and ultrasound examination, and DSA is used as golden reference
  Interventions: Diagnostic Test: 3D-TOF-MRA

INTERVENTIONS:
Diagnostic Test: 3D-TOF-MRA — The Principle of 3D-TOF-MRA is based on the "flow effect" of MR. In the GE sequence of MRA imaging, the effect of RF pulses makes the protons in the stationary tissue in the active layer in a saturated state, and the longitudinal magnetization disappears. When the inflow blood appears, its protons are in an unsaturated state and have a high degree of longitudinal magnetization. In this way, a clear difference is formed between saturated tissue and unsaturated flowing blood to display blood vessels. 3D-TOF-MRA is a non-invasive and safe method for diagnosing vascular diseases.
  Other Names: Ultrasound; Digital Substraction Angiography

SUMMARY:
This study is aimed to assess the value of three-dimensional time-of-flight magnetic resonance angiography (3D-TOF-MRA) in hemodialysis patients with occlusive disease in arteriovenous fistula (AVF). All participants will receive 3D-TOF-MRA and ultrasound to detect the stenosis degree of AVF.

DETAILED DESCRIPTION:
The Principle of 3D-TOF-MRA is based on the "flow effect" of MR. In the GE sequence of MRA imaging, the effect of RF pulses makes the protons in the stationary tissue in the active layer in a saturated state, and the longitudinal magnetization disappears. When the inflow blood appears, its protons are in an unsaturated state and have a high degree of longitudinal magnetization. In this way, a clear difference is formed between saturated tissue and unsaturated flowing blood to display blood vessels. Therefore as a non-invasive and safe method for diagnosing vascular diseases, 3D-TOF-MRA is used widely in cerebrovascular diseases. However, there are currently no studies using 3D-TOF-MRA to diagnose arteriovenous fistula (AVF) stenosis in hemodialysis patients. This project plans to use 3D-TOF-MRA to detect AVF stenosis in hemodialysis patients to provide a safe and effective diagnostic method for patients with end-stage renal failure.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients suspected of occlusive disease in arteriovenous fistula (AVF);
* persistent edema of the limb with the fistula;
* decreased pulse or fremitus in anastomotic astium
* increase in venous pressure; blood flow at the access of less than 200 mL/min;

Exclusion Criteria:

* previous endovascular recanalization with stent or graft placement;
* contraindications to magnetic resonance imaging (MRI) examination;
* platelet(PLT)<60*10^9/L or international normalized ratio (INR)>1.5; 4. important organ function failure or other serious illness; 5. Allergic to antiplatelet drug, anticoagulant drug, anaesthetic drug and contrast material.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
degree of stenosis | immediately after examination finished
  visual grading system: 0 = completely smooth vessel wall;
  1. = <50% stenosis;
  2. = 50%-75% stenosis;
  3. = 75%-99% stenosis;
  4. = occlusion.
stenosis location | immediately after examination finished
  1. = arterial vessel of AVF
  2. = orifice of AVF
  3. = venous vessel of AVF

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Qi Zhu, Dr, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made avaliable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT04312711/Prot_SAP_000.pdf